CLINICAL TRIAL: NCT02719236
Title: Direct Anterior Approach Versus Direct Lateral Approach in Cementless Total Hip Arthroplasty
Brief Title: Direct Anterior Approach Versus Direct Lateral Approach in Total Hip Arthroplasty
Acronym: DAAvsDLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Collaborators: Emergency County Hospital Cluj-Napoca (Unknown)
Responsible Party: Principal Investigator, Dan Viorel Nistor, Dan-Viorel Nistor MD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 517/2015
Record Dates: First submitted 2016-02-12; First posted 2016-03-25 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Coxarthrosis
Keywords: Coxarthrosis; Hip arthroplasty; Direct Anterior Approach; Direct Lateral Approach
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct anterior approach (Active Comparator): Primary total hip arthroplasty using a direct anterior approach
  Interventions: Procedure: direct anterior approach
- Direct lateral approach (Active Comparator): Primary total hip arthroplasty using a direct lateral approach
  Interventions: Procedure: direct lateral approach

INTERVENTIONS:
Procedure: direct anterior approach — The procedure begins by positioning the patient supine on a normal table . Both feet are draped separately to assist with dislocating and proximal femural shaft exposure.The surgical incision begins 2-4 cm lateral to the anterior superior iliac spine of the pelvis . It is then carried distally and laterally for about 8-12 cm. After protecting the lateral femoral cutaneous nerve, the fascia overlying the tensor fascia latae (TFL) is incised, and a plane is then developed between the TFL and sartorius. After coagulating the ascending branch of the lateral femoral circumflex artery, a capsulectomy is performed. Placement of the final acetabular component is facilitated by the use of an offset inserter handle.
  Femoral preparation begins by placing the operative limb in a position of extension, adduction and external rotation to improve the accessibility of the proximal femur.
  Once the final implants are in situ, the hip is reduced and assessed.
  Other Names: modified Smith-Peterson approach
  Arms: Direct anterior approach
Procedure: direct lateral approach — The procedure begins by positioning the patient in the supine decubitus position.
  A longitudinal incision is made extending 3-5 cm proximal and about 5-8 cm distal to the tip of the greater trochanter . The fascia is split at the interval between the TFL and gluteus. The tendon and muscle fibres of the gluteus medius are then visualized and split . The gluteus minimus and joint capsule are split. The surgeon then dislocates the femoral head, and performs a femoral neck osteotomy.
  The acetabulum is prepared .Soft tissue landmarks and reamer positioning relative to the floor are used to verify acetabular version and inclination.
  When preparing the proximal femur, the hip is adducted and externally rotated, with the knee flexed. The femural stem is then press-fitted. Once the final implants are in situ and the hip is reduced, the stability of the construct is assessed.
  Other Names: Hardinge approach
  Arms: Direct lateral approach

SUMMARY:
The purpose of this study is to compare the direct anterior approach and the direct lateral approach in primary total hip arthroplasty, regarding the postoperative function and pain, complications, radiological finds (X-ray), postoperative hemorrhage, markers for muscle damage (i.e creatine kinase (CK), lactate dehydrogenase(LDH/LD) , aspartate aminotransferase(AST), C-reactive protein (CRP),Troponin and Myoglobin) or other clinical outcomes.

DETAILED DESCRIPTION:
This is a prospective randomised controlled clinical trial and follow-up study comparing primary total hip arthroplasty performed either through a direct anterior approach or a lateral approach. At our hospital(i.e. Emergency County Hospital Cluj-Napoca), the lateral transgluteal approach was standard for more than 40 years. Starting 2008,the minimally invasive anterior approach was gradually implemented with the aim to facilitate early rehabilitation and improve functional results. Reduced blood loss, earlier functional recovery, low dislocation rates and shorter stays in hospital have been attributed to the muscle-sparing properties of the anterior approach.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of coxarthrosis
* Those deemed capable of giving informed consent, understanding the aims of the study and expressing willingness to comply with the post-operative review programme.

Exclusion Criteria:

* Previous surgery on affected hip
* The patient has inflammatory arthritis.
* The patient has any type of infection.
* The subject has a known metal allergy.
* Patients with co-existent ipsilateral knee disease or back problems
* Those with a known co-existent medical condition where death is anticipated within five years due to the pre-existing medical condition.
* Patients requiring bilateral hip replacement.
* Patient with active major psychiatric illness
* Patients whose body mass index (BMI; kg/m2) >35.
* Patients with active or suspected infection or sepsis.
* Patients with renal failure and/or renal insufficiency.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-03; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Muscle damage assay using Myoglobin biomarker | Day of surgery
  Before surgery, Myoglobin(ng/mL) baseline value is acquired in the morning, prior to any physical activity. Myoglobin value postoperatively is acquired at the 6 hour mark, when it reaches peak level. The change from baseline of the biomarker is calculated considering patient haemodilution.
Muscle damage assay using Troponin T biomarker | Day of surgery
  Before surgery, Troponin T(pg/mL) baseline value is acquired in the morning ,prior to any physical activity.Troponin T(TnT) value postoperatively is acquired at the 6 hour mark, when it reaches peak level. The change from baseline of the biomarker is calculated considering patient haemodilution.

SECONDARY OUTCOMES:
Functional outcome using Harris Hip Score | preoperative,and at follow-up visits at 6 weeks, 3 months, 6 months, 12 months and 24 months
  The postoperative rate of improvement in functional outcome, measured by the Harris Hip Score (HHS). The HHS was developed to assess the results of hip surgery and is intended to evaluate pain, function, range of motion and absence of deformity, with a range of possible outcomes from 0 to 100(<70 Poor ;70 - 79 Fair; 80-89 Good; 90 -100 Excellent). The objective is to assess the dynamics of patient clinical recovery comparing functional outcome using HHS at predetermined follow-up visits and pre-op.
Functional outcome using the Oxford Hip Score Survey | preoperative,and at follow-up visits at 6 weeks, 3 months, 6 months, 12 months and 24 months
  The Oxford hip score (OHS) is a joint specific outcome measure tool designed to assess disability in patients undergoing total hip replacement (THR).The OHS is a patient-centred questionnaire that is designed to assess functional ability, and pain from the patient's perspective. It is a short, twelve-item questionnaire. Each item has five response categories, given a score of between 1-5 (low disability to high disability). Scoring involves summating the total for each item to produce a final score between 12-60, with a higher score indicating greater disability The objective is to assess the dynamics of patient clinical recovery comparing the OHS at predetermined follow-up visits and pre-op.
Functional outcome using the 36-Item Short Form Health Survey (SF-36) | preoperative,and at follow-up visits at 6 weeks, 3 months, 6 months, 12 months and 24 months
  The SF-36 Survey consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.The eight sections are: vitality,physical, functioning,bodily pain,general health perceptions,physical role functioning,emotional role functioning, social role functioning and mental health.The objective is to assess the dynamics of patient clinical recovery comparing the SF-36 survey at predetermined follow-up visits and pre-op.
Functional outcome using the 20-meters-timed-walk(66 feet) test | at follow-up visits at 6 weeks, 3 months, 6 months, 12 months and 24 months
  Performance-based measures such as the 20 meters timed walk (20MTW) Test quantify performance with tasks mimicking activities of daily living, as opposed to relying on individuals perception of performance.Hence, they may provide a more objective measure of functional capacity. The test consists in timing the patient while walking a distance of 20 meters(66feet).
Functional outcome using the Stair Climbing Test (SCT) | at follow-up visits at 6 weeks, 3 months, 6 months, 12 months and 24 months
  Performance-based measures such as the Stair Climbing Test (SCT) quantify performance with tasks mimicking activities of daily living, as opposed to relying on individuals perception of performance.Hence, they may provide a more objective measure of functional capacity. The test consists in timing the patient while climbing 10 steps.
Post Operative Pain Medication Usage | first 7 postoperative days - on a daily basis and then weekly for a 3 months period
  Postoperative, the amount of analgetics used by each patient is quantified (converted to opioid equivalent doses)
Pain assessment using the Visual Numeric Scale | first 7 postoperative days - on a daily basis and then weekly for a 3 months period
  The pain felt by the patient is measured using the Visual Numeric Scale(VNS) consisting of a scale from 0-10 (0 = no pain; 10 = worst imaginable pain).
Muscle damage - Creatine kinase (CK) | Day of operation and next 7 consecutive days
  Creatine kinase (CK) - also known as creatine phosphokinase (CPK) or phospho-creatine kinase - is an enzyme expressed by various damaged tissues. Baseline value is acquired before surgery.CK-total is measured daily, the first post-op week,in the morning, to avoid physiological circadian variations.
Muscle damage - Lactate dehydrogenase (LDH or LD) | Day of operation and next 7 consecutive days
  Lactate dehydrogenase (LDH or LD) is an enzyme found in nearly all living cells.LDH is expressed extensively in body tissues, such as blood cells and heart muscle. Because it is released during tissue damage, it is a marker of common injuries and disease such as surgical muscle damage. Baseline value is acquired before surgery. LDH is measured daily, the first post-op week,in the morning, to avoid physiological circadian variations.
Muscle damage assay using Aspartate aminotransferase (AST) | Day of operation and next 7 consecutive days
  Aspartate aminotransferase (AST) is found in the liver, heart, skeletal muscle, kidneys, brain, and red blood cells. Serum AST level can be measured clinically as biomarker for muscle health. Baseline value is acquired before surgery. AST is measured daily, the first post-op week,in the morning, to avoid physiological circadian variations.
radiological assessment of cup positioning in the replaced hip | first day postoperative
  Using standard X-ray of the hip - Placement of the acetabular component (inclination and version) is assessed on a Anterior-Posterior view (AP) and a Rolled Lateral view. The outcome measured is correct component placement, within the accepted range.
radiological assessment of stem positioning in the replaced hip | first day postoperative
  Using standard X-ray of the hip , placement of the stem is assessed on a Anterior-Posterior view (AP) and a Rolled Lateral view. The outcome measured is correct component placement, within the accepted range.
radiological assessment of cup and stem osteointegration in the replaced hip | 12 months postoperative
  The outcome measured is correct component osteointegration of the acetabular component and femoral stem using standard X-ray of the replaced hip.
Length of Hospital Stay | 10 days postoperative
  The length of stay will be determined for each patient,to evaluate and compare the percentage of patients who are able to be discharged in less than 5 days after undergoing total hip arthroplasty through either a direct anterior or lateral approach, utilizing the identical post operative protocol for physical recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Dan V Nistor, MD, Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy; Adrian Todor, MD, PhD, Study Director — Iuliu Hatieganu University of Medicine and Pharmacy
Locations (1):
- Emergency County Hospital Cluj-Napoca, Orthopedics and Trauma Clinic, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Matta JM, Shahrdar C, Ferguson T. Single-incision anterior approach for total hip arthroplasty on an orthopaedic table. Clin Orthop Relat Res. 2005 Dec;441:115-24. doi: 10.1097/01.blo.0000194309.70518.cb. PMID 16330993
- [Background] Petis S, Howard JL, Lanting BL, Vasarhelyi EM. Surgical approach in primary total hip arthroplasty: anatomy, technique and clinical outcomes. Can J Surg. 2015 Apr;58(2):128-39. doi: 10.1503/cjs.007214. PMID 25799249
- [Background] Ilchmann T, Gersbach S, Zwicky L, Clauss M. Standard Transgluteal versus Minimal Invasive Anterior Approach in hip Arthroplasty: A Prospective, Consecutive Cohort Study. Orthop Rev (Pavia). 2013 Nov 6;5(4):e31. doi: 10.4081/or.2013.e31. eCollection 2013. PMID 24416475
- [Background] Chechik O, Khashan M, Lador R, Salai M, Amar E. Surgical approach and prosthesis fixation in hip arthroplasty world wide. Arch Orthop Trauma Surg. 2013 Nov;133(11):1595-600. doi: 10.1007/s00402-013-1828-0. Epub 2013 Aug 4. PMID 23912418
- [Background] Connolly KP, Kamath AF. Direct anterior total hip arthroplasty: Literature review of variations in surgical technique. World J Orthop. 2016 Jan 18;7(1):38-43. doi: 10.5312/wjo.v7.i1.38. eCollection 2016 Jan 18. PMID 26807354
- [Background] De Anta-Diaz B, Serralta-Gomis J, Lizaur-Utrilla A, Benavidez E, Lopez-Prats FA. No differences between direct anterior and lateral approach for primary total hip arthroplasty related to muscle damage or functional outcome. Int Orthop. 2016 Oct;40(10):2025-2030. doi: 10.1007/s00264-015-3108-9. Epub 2016 Jan 12. PMID 26753844
- [Background] Dayton MR, Judd DL, Hogan CA, Stevens-Lapsley JE. Performance-Based Versus Self-Reported Outcomes Using the Hip Disability and Osteoarthritis Outcome Score After Total Hip Arthroplasty. Am J Phys Med Rehabil. 2016 Feb;95(2):132-8. doi: 10.1097/PHM.0000000000000357. PMID 26259051
- See also: Romanian Arthroplasty Register — http://www.rne.ro/